CLINICAL TRIAL: NCT04651153
Title: A Multicenter, Participant-Blind, Investigator-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of UCB7853 in Healthy Male Study Participants and Multiple Ascending Doses in Patients With Parkinson's Disease
Brief Title: A Safety and Pharmacokinetics Study of UCB7853 in Healthy Study Participants and Study Participants With Parkinson's Disease (PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0092; 2020-003356-32 (EudraCT Number)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Phase 1; Healthy Volunteers; Patients
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCB7853 (Experimental): Part 1: Single intravenous infusion of UCB7853 Part 2: Multiple intravenous infusions of UCB7853 at pre-specified time-points
  Interventions: Drug: UCB7853
- Placebo (Placebo Comparator): Part 1: Single intravenous infusion of Placebo Part 2: Multiple intravenous infusions of Placebo at pre-specified time-points
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB7853 — Subjects will receive UCB7853 at pre-specified time-points.
  Arms: UCB7853
Other: Placebo — Subjects will receive Placebo at pre-specified time-points.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of single ascending doses of UCB7853 in healthy male study participants and to evaluate the safety and tolerability of multiple ascending doses of UCB7853 administered in study participants with Parkinson's Disease (PD)

ELIGIBILITY:
Inclusion Criteria:

Part 1 (healthy participants):

* Participant must be male and 18 to 55 years of age inclusive
* Body weight within 50 kg to 110 kg and body mass index (BMI) within the range 18.0 to 30.0 kg/m^2 (inclusive)
* Participant must be healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant has clinical laboratory test results within the reference ranges of the laboratory

Part 2 (participants with Parkinson's Disease):

* Participant must be 40 to 80 years of age, inclusive, at the time of signing the informed consent form (ICF)
* Participant may be male or female
* Participant must have body weight of between 50 and 110 kg and a body mass index within the range of 18 to 32 kg/m^2 (inclusive)
* Participant must have a clinical diagnosis of Parkinson's disease (PD) according to the Movement Disorders Society criteria. The following diagnostic criteria must be met: Bradykinesia AND at least ONE of the following: muscular rigidity or resting tremor
* Participant must have a Hoehn and Yahr Stage of ≤3
* Participant must be either untreated, or treated with a stable regimen (at least 4 weeks prior to Baseline Visit) of antiparkinsonian drugs and is expected to remain on this regimen for the duration of the study
* Participant must be in good physical and mental health, in particular not affected by any neurological disorder other than Parkinson's disease (PD), in the opinion of the Investigator, determined on the basis of medical history and a general clinical examination at Screening
* Participant has clinical laboratory test results within the reference ranges of the laboratory

Exclusion Criteria:

Part 1 (healthy participants):

* Participant has a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, pancreatic, musculoskeletal, genitourinary, immunological, dermatological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs
* Participant has any clinically relevant abnormal findings in physical examination, laboratory tests, or vital signs, which, in the opinion of the Investigator, may place the participant at risk because of participation in the study
* Participant has any clinically relevant brain magnetic resonance imaging (MRI) abnormality at Screening

Part 2 (participants with Parkinson's Disease):

* Participant has a diagnosis of a significant Central nervous system (CNS) disease other than PD or history of epilepsy or seizure disorder other than febrile seizures as a child
* Study participant has a history of levodopa-induced motor fluctuations or dyskinesia expected to interfere with his/her ability to participate in the study
* Participant has a known hypersensitivity to any components of the study medication or comparative drugs
* Study participant has had prior surgical treatment for PD involving intracranial surgery or implantation of a device (including deep brain stimulation) or duodopa
* Participant has any clinically relevant abnormal findings in physical examination (other than symptoms of PD), laboratory tests, or vital signs, which, in the opinion of the Investigator, may place the participant at risk because of participation in the study
* Participant has any clinically relevant brain MRI abnormality at Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) in healthy male participants | From Day 1 to the End of Study Visit (Day 141), Part 1)
  A treatment-emergent Adverse Event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.
Incidence of Treatment-emergent Adverse Events (TEAEs) in participants with Parkinson's Disease | From Day 1 to the End of Study Visit (Day 197), Part 2
  A treatment-emergent Adverse Event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.

SECONDARY OUTCOMES:
Cmax of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from Day 1 to the End of Study Visit (Day 141), Part 1
  Cmax = Maximum observed concentration
Cmax of UCB7853 in serum after intravenous infusion of multiple ascending doses in study participants with Parkinson's Disease | Samples will be taken from Day 57 to the End of Study Visit (Day 197), Part 2
  Cmax = Maximum observed concentration
AUC of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from Day 1 to the End of Study Visit (Day 141), Part 1
  AUC = Area under the concentration-time curve
AUC(0-t) of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from Day 1 to the End of Study Visit (Day 141), Part 1
  AUC(0-t) = Area under the concentration-time curve from time 0 to time t
AUC(0-t) of UCB7853 in serum after intravenous infusion of multiple ascending doses in study participants with Parkinson's Disease | Samples will be taken from Day 57 to Day 85, Part 2
  AUC(0-t) = Area under the concentration-time curve from time 0 to time t
tmax of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from Day 1 to the End of Study Visit (Day 141), Part 1
  tmax = Time to reach Cmax
tmax of UCB7853 in serum after intravenous infusion of multiple ascending doses in study participants with Parkinson's Disease | Samples will be taken from from Day 57 to the End of Study Visit (Day 197), Part 2
  tmax = Time to reach Cmax
t1/2 of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from Day 1 to the End of Study Visit (Day 141), Part 1
  t1/2 = Terminal half-life
CL of UCB7853 after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from from Day 1 to the End of Study Visit (Day 141), Part 1
  CL = Total body clearance of the drug
CL of UCB7853 after intravenous infusion of multiple ascending doses in study participants with Parkinson's Disease | Samples will be taken from from Day 57 to Day 85, Part 2
  CL = Total body clearance of the drug
Vz of UCB7853 in serum after intravenous infusion of single ascending doses in healthy male participants | Samples will be taken from from Day 1 to the End of Study Visit (Day 141), Part 1
  Vz = Volume of distribution during terminal phase
CSF/serum UCB7853 concentration ratio on Day 7 (Part 1) | Day 7 (Part 1)
  CSF = Cerebrospinal fluid
CSF/serum UCB7853 concentration ratio on Day 63 (Part 2) | Day 63 (Part 2)
  CSF = Cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (2):
- Up0092 201, Leiden, Netherlands
- Up0092 101, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.